CLINICAL TRIAL: NCT01834625
Title: Prognostic Value of Aβ Imaging in NPH Prior to Shunt Placement
Status: Terminated | Type: Observational
Why Stopped: not recruiting
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Neill R. Graff-Radford, M.D., Professor of Neurology, Mayo Clinic
Other Study IDs: 11-004532
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2018-02

CONDITIONS: Normal Pressure Hydrocephalus Patients
MeSH Terms: interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Florbetapir +ve NPH patients: Florbetapir +ve patients will have neuropsychology tests prior to surgery and then at 3 and 12 months
  Interventions: Diagnostic Test: PET scan
- Florbetapir -ve patients: Florbetapir -ve patients will have neuropsychology tests prior to surgery and then at 3 and 12 months
  Interventions: Diagnostic Test: PET scan

INTERVENTIONS:
Diagnostic Test: PET scan

SUMMARY:
In this pilot study the investigators shall prospectively in a blinded fashion evaluate with Aβ PET in patients committed to shunt surgery and then investigate the relationship of these biomarkers with outcome on gait, cognition and urinary control improvement in the short term (3 months) and long term (1 year). The imaging agent will be provided by AVID.

Furthermore the study will standardize imaging studies using florbetapir F 18 PET to provide information on amyloid burden.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60.
2. Visual and auditory acuity adequate for neuropsychological testing.
3. Completed six grades of education or has a good work history (sufficient to exclude mental retardation).
4. Must speak English fluently.
5. Willing to undergo one Amyloid imaging PET scan.
6. Agrees to at least one lumbar puncture for the collection of CSF.
7. Must agree to return for a Month 3 and Month 12 visit.
8. Participant, who in the opinion of the investigator, can tolerate the PET scan procedures

Exclusion Criteria:

1. History of schizophrenia (DSM IV criteria).
2. History of alcohol or substance abuse or dependence within the past 2 years (DSM IV criteria).
3. Participation in clinical studies involving neuropsychological measures being collected more than one time per year.
4. Exclusion for amyloid imaging with 18F -AV-45: Current or recent participation in any procedures involving radioactive agents such that the total radiation dose exposure to the participant in any given year would exceed the limits of annual and total dose commitment set forth in the US Code of Federal Regulations (CFR) Title 21 Section 361.1.
5. Clinically significant hepatic, renal, pulmonary, metabolic, or endocrine disturbances as indicated by history, which in the opinion of the investigator might pose a potential safety risk to the participant?
6. Current clinically significant cardiovascular disease, including one or more of:

   * cardiac surgery or myocardial infarction within the last 4 weeks;
   * unstable angina;
   * acute decompensated congestive heart failure or class IV heart failure

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically evaluated NPH patients
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2013-04; Primary Completion 2017-03 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Comparison of change between florbetapir +ve and -ve patients from baseline to one year in the Montreal Cognitive Assessment (MoCA) | Baseline to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Neill R Graff-Radford, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States